CLINICAL TRIAL: NCT06501014
Title: Investigating the Effectiveness of Action Observation Therapy Applied in Addition to Conventional Treatment in Stroke Patients
Brief Title: Effectiveness of Action Observation Therapy in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUO3
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy-Experimental Group (Experimental): Patients will be asked to watch the exercises before doing them. For each exercise, patients will first watch the relevant video and do the exercise after the video ends.
  Interventions: Other: Action Observation Therapy-Experimental Group
- Conventional Exercises-Control Group (Active Comparator): Patients will be subjected to conventional exercise only.
  Interventions: Other: Conventional Exercises-Control Group

INTERVENTIONS:
Other: Action Observation Therapy-Experimental Group — Patients will be asked to watch the exercises before doing them.For each exercise, patients will first watch the relevant video and do the exercise after the video ends.
  Arms: Action Observation Therapy-Experimental Group
Other: Conventional Exercises-Control Group — Patients will be subjected to conventional exercise only.
  Arms: Conventional Exercises-Control Group

SUMMARY:
The goal of this clinical trial is to learn the effectiveness of action observation therapy in patients with stroke.

The main questions it aims to answer are:

Is action observation therapy an effective method in stroke patients?

Researchers will compare the results of two action observation-based exercises (home program) with conventional exercise to see whether action observation therapy works in the rehabilitation of stroke patients.

Participants:

Participants in one group will do action observation-based exercise (home plus conventional exercise for 24 sessions, Patients in the control group will only undergo conventional exercise in addition to routine treatment.

DETAILED DESCRIPTION:
Individuals with chronic stroke will be included in this study. Participants will be randomly divided into two groups, and patients in both groups will continue their routine treatments.

Patients in the control group will only undergo conventional exercise. Patients in the study group will be given a home exercise program in addition to conventional treatment. However, patients will be asked to first watch the video of each exercise in this program and then perform the exercise.

Patients will be asked to perform the exercises 3 days a week for 8 weeks. Evaluations will be made twice, before the exercise program application begins and after the sessions are completed.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients in the chronic phase (more than 6 months have passed since the stroke)
* Patients over 40 years of age
* Patients who can stand and walk independently (including those using walking aids)

Exclusion Criteria:

* Additional disease (neurological, orthopedic, etc.) that may affect motor performance and balance.
* Patients with communication problems
* Patients with mental problems (mini-mental test score <23)
* Patients aged 85 and over

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
2 minute walk test | The evaluation will be applied at the baseline and after study completion, an average of 2 months.
  Patients will be asked to walk 30 meters long on a flat surface for 2 minutes. When the time is up, the distance the patient can walk will be recorded.
Fugl-Meyer Assessment | The evaluation will be applied at the baseline and after study completion, an average of 2 months.
  The FMA motor assessments for the lower extremity (minimum score:0 and maximum score 34 points) will be applied. A higher score means the patient's motor movements are better.
Berg Balance Scale | The evaluation will be applied at the baseline and after study completion, an average of 2 months.
  The Berg Balance Scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of funcion.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Karaca, PhD, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No